CLINICAL TRIAL: NCT02584231
Title: Pharmacokinetics and Pharmacodynamics of Desmopressin Oral Lyophilisate Formulation in the Paediatric Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Principal Investigator, Pediatrie, Prof Johan Vande Walle, University Hospital, Ghent
Organization: University Hospital, Ghent (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EC/2015/0616; 2014-005200-13 (EudraCT Number)
Record Dates: First submitted 2015-09-10; First posted 2015-10-22 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Monosymptomatic Nocturnal Enuresis
Keywords: Desmopressin; Paediatrics; urinary concentration test
MeSH Terms: interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients needing an urinary concentration test (Experimental): Patients who need a urinary concentration test because of uro- or nephropathy (age: 6 months - 8 year)
  Interventions: Drug: desmopressin
- Patients suffering from treatment resistant nocturnal enuresis (Experimental): Patients suffering from treatment resistant nocturnal enuresis (age: 5 - 8 year)
  Interventions: Drug: desmopressin

INTERVENTIONS:
Drug: desmopressin — One time dosing of desmopressin oral lyophilisate formulation. The dose is age-dependant: >6 months and < 2years: 60µg; ≥2 years and <4 years: 120µg PO and ≥4 years and <8 years: 240 µg PO. There will be blood sampling and urine sampling for PK and PD/safety
  Other Names: dDAVP

SUMMARY:
Patients suffering from nocturnal enuresis (starting from the age of 5 till adulthood) are all treated with the same dose of desmopressin, i.e. 120mcg once daily. In treatment resistant enuresis, this dose is doubled: those patients take 240mcg once daily. A pilot study performed at our department showed a correlation between weight and plasma concentration when a fixed dose of desmopressin oral lyophilisate formulation was given to the pediatric patient (older than 6 years). This study will investigate the pharmacokinetics (PK) and pharmacodynamics (PD) of desmopressin in young children, less than 8 years old. Additionally, the efficacy of desmopressin oral lyophilisate formulation in urinary concentration testing will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Children with an uro- and/or nephropathy who need an urinary concentration test OR Children with monosymptomatic nocturnal enuresis (based on nocturnal polyuria) with treatment failure on desmopressin tablet
* Otherwise healthy children (on medical history and physical examination)
* Parents or legal guardian of the child signed the informed consent form
* Age: between 6 months and 8 years
* Minimum weight: 8 kg

Exclusion Criteria:

* Diabetes insipidus
* Renal failure (eGFR<60ml/min/1,73m²)
* Current urinary tract infection
* Syndrome of inappropriate antidiuretic hormone secretion
* Heart failure
* Clinical significant medical conditions (renal, hepatic, gastro-intestinal, pulmonary, cardiac, endocrinologic) that might interfere with the clinical endpoints
* Sensitivity to desmopressin or excipients of the oral lyophilisate formulation
* Use of antibiotics, diuretics or other drugs that can influence diuresis (tricyclic antidepressants, chlorpropamide, oxcarbazepine, selective serotonin reuptake inhibitors, chlorpromazine and carbamazepine).
* Use of drugs that influence intestinal motility (such as loperamide)
* Anomalies of the mouth that might interfere with the intake / absorption of the medication

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Desmopressine concentrations | 24 hours
  The assessed pharmacokinetic parameters are desmopressine concentrations at timepoints 0, 1/4, 1/2, 1, 2, 3, 5, 6 and 7h.

SECONDARY OUTCOMES:
Efficacy - urinary volume. | 24 hours
  PD of desmopressin in children with nocturnal enuresis that is resistant to treatment with desmopressin tablet. First PD parameter is antidiuretic effect. This is urinary volume per hour.
Efficacy - osmolality in urine. | 24 hours
  PD of desmopressin in children with nocturnal enuresis that is resistant to treatment with desmopressin tablet. Second PD parameter is urinary concentration capacity. This is osmolality in urine.
Urinary concentration test | 24 hours
  Evaluation of the oral lyophilisate formulation of desmopressin for the urinary concentration test. Assessed parameter is urinary concentration capacity.
Safety of desmopressin in children as assessed by registration of adverse events. | 24 hours
  Registration of adverse events
Safety of desmopressin in children as assessed by the measurement of natremia. | 24 hours
  Measurement of natremia

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital - Department of Paediatric Nephrology, Ghent, Belgium

REFERENCES:
- [Derived] Michelet R, Dossche L, Van Herzeele C, De Bruyne P, Gasthuys E, Van Bocxlaer J, Vande Walle J, Vermeulen A. An Integrated Paediatric Population PK/PD Analysis of dDAVP: How do PK Differences Translate to Clinical Outcomes? Clin Pharmacokinet. 2020 Jan;59(1):81-96. doi: 10.1007/s40262-019-00798-6. PMID 31347012